CLINICAL TRIAL: NCT04265274
Title: Phase II Study of Vinorelbine, Cisplatin, Disulfiram and Copper in CTC_EMT Positive Refractory Metastatic Breast Cancer.
Brief Title: Vinorelbine, Cisplatin, Disulfiram and Copper in CTC_EMT Positive Refractory Metastatic Breast Cancer.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor acrual
Sponsor: National Cancer Institute, Slovakia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREAST-SK-001
Record Dates: First submitted 2020-02-05; First posted 2020-02-11 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer, vinorelbin, cisplatin, disulfiram
MeSH Terms: conditions — Breast Neoplasms | interventions — Disulfiram; Vinorelbine; Cisplatin; Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disulfiram, vinorelbin, cisplatin, copper (Experimental): Vinorelbine 25mg/m2 day 1 and 8, Cisplatin 75mg/m2 day 1, every 3 weeks, Disulifiram um 400mg daily and 2 mg of elementary Copper daily, continuously.
  Interventions: Drug: Disulfiram; Drug: Vinorelbin; Drug: Cisplatin; Drug: Copper

INTERVENTIONS:
Drug: Disulfiram — dosing 400mg daily
  Other Names: Antabus
Drug: Vinorelbin — 25mg/m2 day 1 and 8,
  Other Names: Navelbine
Drug: Cisplatin — 75mg/m2 day 1
Drug: Copper — 2 mg of elementary Copper daily

SUMMARY:
This is a proof-of-concept study to define efficacy of vinorelbine, cisplatin, disulfiram and copper in CTC_EMT positive refractory metastatic hormone receptor positive, HER2 negative breast cancer.

DETAILED DESCRIPTION:
Despite advances in breast cancer prevention, diagnosis, and therapy, 5-10% of patients with breast cancer have metastatic disease at initial presentation, and approximately 30% of patients with breast cancer develop metastatic disease during the course of disease. Metastatic cascade is a multistep process that enables the migration of tumor cells from the primary site to a distant location, where they can potentially establish a new cancer growth. To execute the metastatic cascade, epithelial cancer cells must detach from the primary tumor, pass through the peripheral circulation, extravasate at the distant site and create a new tumor.

Experimental and clinical data suggest a close relationship between activation of EMT program and generation of CTCs. EMT is associated with a set of molecular changes in epithelial cancer cells that results in increased motility and the induction of proteases that are involved in degradation of the extracellular matrix facilitating thus invasion and intravasation into the bloodstream. EMT has also been linked to the stem cell phenotype and resistance to apoptotic signals, facilitating EMT-derived CTCs to survive in foreign environments. Cancer stem cell phenotype is closely related to ALDH expression. Several studies showed that CTCs with EMT phenotype is associated with inferior outcome in primary as well as in metastatic setting.

In a biomarker study in primary breast cancer, CTC_EMT were detected in 77 (18.0%) of patients. Patients without detectable CTC_EMT in the peripheral blood had significantly superior DFS compared to patients with detectable CTC_EMT (HR = 0.42, 95%CI 0.22 - 0.78, p = 0.0003). Prognostic value of CTC_EMT was demonstrated in all subgroups of patients, most pronounced in hormone receptor positive, HER2 negative subgroup. In multivariate analysis, presence of CTC_EMT, axillary nodal involvement and hormone receptor status were independently associated with DFS. Presence of CTC_EMT could lead to better identification of patients with increased risk of recurrence, especially in hormone receptor positive, HER-2 negative primary breast cancer patients.

Disulfiram (DSF) in combination with copper (Cu) has been reported to override drug resistance in cancer cells, and DSF combined with chemotherapy based on the microtubule inhibitor vinorelbine appears to prolong survival in non-small cell lung cancer patients.

Based on aforementioned data, it is suggested that there is strong rationale to inhibit ALDH in MBC. Inactivation of ALDH by disulfiram/copper will be lead to increase of objective response rate in patients with refractory MBC.

ELIGIBILITY:
Inclusion Criteria:1) Female patients with histologically confirmed carcinoma of the breast.

2) CTC_EMT positivity in the peripheral blood. 3) Patients with locally recurrent or metastatic disease hormone receptor positive, HER2 negative, who have received at least two (and not more than five) prior chemotherapeutic regimens for breast cancer, at least two of which were administered for treatment of locally recurrent and/or metastatic disease.

4) Prior therapy must be documented by the following criteria prior to entry onto study:

* Regimens must have included an anthracycline (e.g., doxorubicin, epirubicin) and a taxane (e.g., paclitaxel, docetaxel) in any combination or order. Treatment with any of these agents is not required if they are contraindicated for a certain patient.
* One or two of these regimens may have been administered as adjuvant and/or neoadjuvant therapy, but at least 2 must have been given for relapsed or metastatic disease.
* Patients must have proved refractory to the most recent chemotherapy, documented by progression on or within six (6) months of therapy.

  5) Patients may have additionally been treated with anti-hormonal therapy. 6) Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy <= Grade 2 and alopecia.

  7) Age >= 18 years. 8) Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2. 9) Life expectancy of >= 3 months. 10) Adequate renal function as evidenced by calculated creatinine clearance >= 40 mL/min per the Cockcroft and Gault formula.

  11) Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >= 1.5 x 10^9/L, hemoglobin >= 9.0 g/dL (a hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion), and platelet count >= 100 x 10^9/L.

  12) Adequate liver function as evidenced by bilirubin <= 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 3 x ULN (in the case of liver metastases <= 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase. In case alkaline phosphatase is >3 x ULN (in absence of liver metastases) or > 5 x ULN (in presence of liver metastases) AND patient is known to have bone metastases, the liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.

  13) Patients willing and able to comply with the study protocol for the duration of the study.

  14) Written informed consent prior to any study-specific screening procedures with theunderstanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received any of the following treatments within the specified period before study treatment start: chemotherapy, radiation, trastuzumab or hormonal therapy within three weeks, any investigational drug within four weeks, radiation therapy encompassing > 30% of marrow.
2. Addiction to alcohol or drugs.
3. Need for metronidazole, warfarin and/or theophylline medication, the metabolism of which is likely influenced by disulfiram and copper, see Table 4.
4. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives, see Table 4.
5. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
6. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g., radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment; radiographic stability should be determined by comparing a contrast-enhanced computed tomography or magnetic resonance imaging brain scan performed during screening to a prior scan performed at least 4 weeks earlier.
7. Patients with meningeal carcinomatosis.
8. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
9. Severe/uncontrolled intercurrent illness/infection.
10. Patients with organ allografts requiring immunosuppression.
11. Patients with known positive HIV status.
12. Hemochromatosis.
13. Patients who have had a prior malignancy, other than previous breast cancer, carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated >= 5 years previously with no subsequent evidence of recurrence.
14. Patients with pre-existing neuropathy > Grade 2.
15. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Objective response rates | 6 months
  Response rate according to RECIST

SECONDARY OUTCOMES:
Progression-free survival | 12 months
  Time from first administration of the study drug till progression
overall survival | 12 months
  Time from first administration of the study drug till death

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, Prof, Study Chair — National Cancer Institute, Slovakia
Locations (1):
- National Cancer Institute, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No